CLINICAL TRIAL: NCT05162625
Title: Safety and Efficacy of Topical Moxifloxacin for Prevention of Post-Traumatic Endophthalmitis: Randomized Controlled Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Mathias Violante Mélega, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 52246021.8.0000.5404
Record Dates: First submitted 2021-11-23; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Endophthalmitis; Open Globe Injury; Moxifloxacin; Post-Traumatic Endophthalmitis
MeSH Terms: conditions — Endophthalmitis | interventions — Ophthalmic Solutions; Ciprofloxacin; Cefazolin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Moxifloxacin (Active Comparator): Pre-surgical prophylaxis with the use of topical 0.5% moxifloxacin eye drops every 3 hours until the surgery.
  Interventions: Drug: Moxifloxacin Ophthalmic 0.5% Ophthalmic Solution
- Intravenous Cephazolin and Ciprofloxacin (Active Comparator): Pre-surgical prophylaxis with cefazolin 1 gram every 6 hours and ciprofloxacin 400 milligrams intravenously every 12 hours, until the surgery.
  Interventions: Drug: Ciprofloxacin 400 MG/200 ML Intravenous Solution [CIPRO IV]

INTERVENTIONS:
Drug: Moxifloxacin Ophthalmic 0.5% Ophthalmic Solution — Topical moxifloxacin 0,5% 01 drop every 3 hours
  Arms: Topical Moxifloxacin
Drug: Ciprofloxacin 400 MG/200 ML Intravenous Solution [CIPRO IV] — Intravenous ciprofloxacin 400mg every 12 hours and cefazolin 1000mg every 6 hours
  Other Names: + Cefazolin
  Arms: Intravenous Cephazolin and Ciprofloxacin

SUMMARY:
Open globe injuries (OGI) are among the main causes of blindness or irreversible severe reduction in visual acuity in the world. An estimated 2.3 million people live with bilateral low vision and nearly 19 million live with blindness or unilateral low vision due to such trauma. Pre-surgical prophylaxis to prevent serious infectious complications such as endophthalmitis is frequently performed, however, there are discrepancies in its performance between services as there is no proven superior protocol. Different combinations of antibiotics and administration routes are currently used.

The aim of this study is to evaluate the efficacy and safety of the use of topical moxifloxacin 0.5% ophthalmic solution (Vigamox®) in the prophylaxis of acute endophthalmitis in patients with OGI. This is a prospective, controlled, randomized, single-center study conducted in patients diagnosed with OGI at the Clinical Hospital of São Paulo State University, Campinas.

Volunteers who present OGI and sign the informed consent form (ICF) will be randomized into 2 groups: in group A, volunteers will undergo pre-surgical prophylaxis with the use of topical 0.5% moxifloxacin eye drops every 3 hours until the surgery.

In group B, the volunteers will receive pre-surgical prophylaxis as it is currently done in the service, with cefazolin 1 gram every 6 hours and ciprofloxacin 400 milligrams intravenously every 12 hours, prior to surgery. Intraoperative and post-surgical care will be the same for both groups and will continue to be carried out in line with the current service protocol. Patients will be followed for 45 days, with a complete ophthalmological evaluation that aims to verify the incidence of endophthalmitis in both groups. It is expected to find an equal or lower incidence of endophthalmitis in the group that received topical administration of moxifloxacin.

DETAILED DESCRIPTION:
Patients diagnosed with OGI that requires surgery will be evaluated regarding visual acuity, biomicroscopy and fundoscopy, considering that the latter may not be possible in some cases due to the trauma severity. Those who, after being informed about all aspects of the surgery and this study, sign the ICF will be randomly divided into 2 groups of approximately equal sizes stratified by gender. Group A will receive, throughout the preoperative period, instillation of 0.5% moxifloxacin eye drops, 01 drop every 3 hours until the time of surgery. Group B will receive intravenous use of cefazolin 1 gram every 6 hours and ciprofloxacin 400mg every 12 hours.

The primary outcome is to evaluate the incidence of endophthalmitis in each group. The secondary outcome is to assess the other possible postoperative complications such as corneal decompensation and development of glaucoma and cataract, as well as analysis of the epidemiological profile of patients.

All patients will be hospitalized throughout the preoperative period, waiting for urgent surgery. All patients will remain with a non-compressive occlusive dressing during the preoperative period, being removed intraoperatively. The dressing will be removed and replaced only for the instillation of eye drops in patients allocated to group A. The surgery to correct OGI will be performed as already standardized in the Ophthalmology service at UNICAMP, by residents of the 3rd and 4th years, as well as assistant physicians and professors for cases of greater complexity and supervising all surgical procedures. The anesthetic technique will be performed according to the current protocol with general anesthesia. Skin antisepsis will be done with 10% aqueous povidone-iodine solution and then sterile surgical drapes will be placed with the eyelashes isolated.

The surgical technique will vary according to the trauma mechanism and the degree of ocular involvement, being defined by the preoperative surgical indication, but it may undergo changes according to the intraoperative evaluation.

Patients in both groups who present involvement of the lens and require its removal during surgery (facectomy) will receive an injection of 0.03ml of 0.5% moxifloxacin intracameral at the end of the surgery, as already standardized in the hospital. For the other cases, in which the lens is not affected, there will be no intracameral injection of 0.5% moxifloxacin.

All patients will receive instillation of 0.5% moxifloxacin eye drops associated with 0.1% dexamethasone (Vigadexa®) after the end of surgery and before the occlusive dressing. The postoperative prescription will consist of 0.5% moxifloxacin associated with 0.1% dexamethasone starting 3 hours after the end of the surgery, at a frequency of every 3 hours until the time the patient goes to sleep, for 7 days. After the 7th day Vigadexa® will be replaced by 0.1% dexamethasone without association with moxifloxacin and will be regressed weekly according to the inflammatory response of each individual.

Patients in both groups will not be masked as they will know if they are receiving eye drops or intravenous medication. Surgeons and ophthalmologists who will perform the exam in the postoperative period will not be masked.

In case of suspected endophthalmitis, an independent ophthalmologist of the retina and vitreous service will assess the patient, without knowing whether he belongs to group A or B, and will indicate the most appropriate procedure. The treatment of endophthalmitis will follow the hospital protocol. Postoperative consultations will take place on the 1st, 7th, 30th and 45th postoperative days with assessment of visual acuity (7th, 30th, 45th), refraction (30th), biomicroscopy (1st, 7th, 45th), tonometry of applanation (7th, 30th and 45th), keratometry (30th) funduscopy (30th and 45th), and endothelial cell count (45th). Occasionally, the performance of some of the aforementioned exams can be impaired by the ocular alteration resulting from OGI.

ELIGIBILITY:
Inclusion Criteria:

* Open globe injury

Exclusion Criteria:

* Under 18 years old
* Requires intravenous antibiotics for other reasons
* Moxifloxacin allergy
* Imunossupressed patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants that develop post-traumatic acute endophthalmitis in each group as assessed by a retina specialist according to clinical exam and ultrasonography findings | Will be considered post-traumatic acute endophthalmitis if the patient evolve the condition until 45 days after open globe injury surgery
  Post-traumatic endophthalmitis incidence rate in each group ( group A: topical moxifloxacin and group B: intravenous cefazolin plus ciprofloxacin)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, Campinas, Brazil